CLINICAL TRIAL: NCT04269226
Title: The Effect of Automatic Recruitment Maneuver on Peroperative Lung Mechanics and Postoperative Kidney Functions of Obese Patients Undergoing Laparoscopic Abdominal Surgery
Brief Title: Effect of Automatic Recruitment Maneuver on Peroperative Lung Mechanics of Obese Laparoscopic Abdominal Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20190409
Record Dates: First submitted 2020-02-09; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Recruitment; Obesity, Morbid; Laparoscopy
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recruitment maneuver (Experimental): Recruitment maneuver
  Interventions: Procedure: Recruitment maneuver
- No recruitment maneuver (Active Comparator): No recruitment maneuver
  Interventions: Procedure: No recruitment maneuver

INTERVENTIONS:
Procedure: Recruitment maneuver — Following intubation, patients will be ventilated according to the ideal weight within the scope of intraoperative protective ventilation strategy and in pressure-controlled ventilation (PCV) mode. Then, automatic recruitment maneuver will be applied to the recruitment group twice, after insufflation and desufflation. It will not be applied to the control group. During recruitment maneuver, PEEP (Positive end-expiratory pressure), where dynamic compliance is measured highest, will be the ideal peep for the patient, and PEEP will be adjusted at this value after recruitment.
  Arms: Recruitment maneuver
Procedure: No recruitment maneuver — Usual ventilation procedures will be applied.
  Arms: No recruitment maneuver

SUMMARY:
This study aims to demonstrate the effects of automatic recruitment maneuver on peroperative lung mechanics of obese patients undergoing laparoscopic abdominal surgery.

128 obese patients undergoing abdominal laparoscopic surgery are randomly going to be assigned to automatic recruitment maneuver group and no recruitment maneuver group (control group). Both groups are going to be taken to the operating table. Electrocardiography (ECG), noninvasive blood pressure (NIBP), pulse oximeter and peripheral oxygen saturation (SpO2) and post-intubation end-tidal carbon dioxide (EtCO2) and train of four (TOF) monitoring will be performed. Then, general anesthesia induction procedure will be started. Following intubation, patients will be ventilated according to the ideal weight within the scope of intraoperative protective ventilation strategy and in pressure-controlled ventilation (PCV) mode. Then, automatic recruitment maneuver will be applied to the recruitment group twice, after insufflation and desufflation. It will not be applied to the control group. During recruitment maneuver, PEEP (Positive end-expiratory pressure), where dynamic compliance is measured highest, will be the ideal PEEP (Positive end-expiratory pressure) for the patient, and PEEP (Positive end-expiratory pressure) will be adjusted at this value after recruitment. If MAP (mean arterial pressure) is <60 mmHg during the maneuver, the maneuver will be terminated and these patients will be excluded from the study. Respiratory mechanics for both groups (peak pressure, plateau pressure, driver pressure, static compliance, dynamic compliance, EtCO2) and hemodynamic parameters (heart peak, mean arterial pressure, SpO2) at 5 different times (T1: post intubation; T2 : after insufflation; T3: 5 minutes after insufflation / after the first recruitment maneuver; T4: after desufflation; T5: 5 minutes after desufflation / after the second recruitment maneuver) will be recorded. Throughout the surgery, insufflation pressure will be kept as 10-13 cmH20. At the end of the surgery, the anesthesia maintenance of all patients will be terminated and the routine wake-up phase will be initiated. Creatinine values and hourly urine outputs of all patients routinely monitored at the postoperative 24th hour will be recorded on the case follow-up form.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18 and 65
2. Body mass index (BMI)> 30 patients undergoing laparoscopic abdominal surgery
3. ASA (American Society of Anesthesiologists) 2-3 patients

Exclusion Criteria:

1. Smokers
2. Patients with previous abdominal surgery
3. Patients with obstructive / restrictive lung disease,
4. Patients with coronary artery disease, heart failure
5. Patients with chronic kidney failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-04-09 (Estimated); Study Completion 2020-05-09 (Estimated)

PRIMARY OUTCOMES:
Peak airway pressure | 1 week
  This will me measured at 5 different times using mechanic ventilator and will be reported as mmHg(T1: post intubation; T2: post insufflation; T3 : 5 minutes after insufflation / after the first recruitment maneuver; T4: after desufflation; T5: 5 minutes after desufflation / after the second recruitment maneuver)
Plateau airway pressure | 1 week
  This will me measured at 5 different times using mechanic ventilator and will be reported as mmHg(T1: post intubation; T2: post insufflation; T3 : 5 minutes after insufflation / after the first recruitment maneuver; T4: after desufflation; T5: 5 minutes after desufflation / after the second recruitment maneuver)
Driver airway pressure | 1 week
  This will me measured at 5 different times using mechanic ventilator and will be reported as mmHg (T1: post intubation; T2: post insufflation; T3 : 5 minutes after insufflation / after the first recruitment maneuver; T4: after desufflation; T5: 5 minutes after desufflation / after the second recruitment maneuver)
Static airway compliance | 1 week
  This will me measured at 5 different times using mechanic ventilator and will be reported as This will me measured at 5 different times using mechanic ventilator and will be reported as cmH2O (T1: post intubation; T2: post insufflation; T3 : 5 minutes after insufflation / after the first recruitment maneuver; T4: after desufflation; T5: 5 minutes after desufflation / after the second recruitment maneuver)
Dynamic airway compliance | 1 week
  This will me measured at 5 different times using mechanic ventilator and will be reported as This will me measured at 5 different times using mechanic ventilator and will be reported as cmH2O (T1: post intubation; T2: post insufflation; T3 : 5 minutes after insufflation / after the first recruitment maneuver; T4: after desufflation; T5: 5 minutes after desufflation / after the second recruitment maneuver)
End tidal CO2 pressure | 1 week
  This will me measured at 5 different times using mechanic ventilator and will be reported as mmHg (T1: post intubation; T2: post insufflation; T3 : 5 minutes after insufflation / after the first recruitment maneuver; T4: after desufflation; T5: 5 minutes after desufflation / after the second recruitment maneuver)

SECONDARY OUTCOMES:
Heart rate | 1 week
  This will me measured at 5 different times using electrocardiography and will be reported as beat per minute (T1: post intubation; T2: post insufflation; T3 : 5 minutes after insufflation / after the first recruitment maneuver; T4: after desufflation; T5: 5 minutes after desufflation / after the second recruitment maneuver)
Mean arterial pressure | 1 week
  This will me measured at 5 different times using non invasive blood pressure monitor and will be reported as mmHg (T1: post intubation; T2: post insufflation; T3 : 5 minutes after insufflation / after the first recruitment maneuver; T4: after desufflation; T5: 5 minutes after desufflation / after the second recruitment maneuver)
SpO2 | 1 week
  SpO2 will me measured at 5 different times using pulse oximetry and will be reported as mmHg (T1: post intubation; T2: post insufflation; T3 : 5 minutes after insufflation / after the first recruitment maneuver; T4: after desufflation; T5: 5 minutes after desufflation / after the second recruitment maneuver)
Creatinine | 24th hour
  Creatinine values will be measured at 24th our using blood tests and will be reported as mg/dL
Urine output | 24th hour
  This will be measured hourly for the first 24 hours, using urinary catheter and will be reported as ml per hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No